CLINICAL TRIAL: NCT06272513
Title: Exploring Influencing Factors for Physical Activity Participation in People With Advanced Head and Neck Cancer - a Qualitative Study
Brief Title: Influencing Factors for Physical Activity in People With Head and Neck Cancer
Acronym: ProAct-HNC
Status: Completed | Type: Observational
Sponsor: Kantonsspital Winterthur KSW (Other)
Collaborators: Eastern Switzerland University of Applied Sciences (Other); University of Applied Sciences of Western Switzerland (Other); UMC Utrecht (Other); University of Lausanne (Other); Zurich University of Applied Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: ProAct-HNC-02
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Advanced Head and Neck Squamous Cell Carcinoma
Keywords: qualitative research; interviews; focus groups; physical activity; health promotion
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this qualitative study is to explore influencing factors for physical activity (PA) participation in people affected by an advanced head and neck cancer from the perspective of people affected and their significant others.

Individual interviews will be conducted with people affected by head and neck cancer and focus group interviews will be held with significant others of people being affected to answer the following research questions:

* What capabilities and opportunities for physical activity participation do people with advanced head and neck cancer experience?
* What motivates people with advanced head and neck cancer to be physically active?
* What are recommendations and suggestions for a future physical activity promotion intervention?
* How do significant others view capabilities, opportunities, and motivation for physical activity participation and promotion in people with head and neck cancer?

The interviews will be transcribed verbatim and analysed with a structuring content analysis approach.

DETAILED DESCRIPTION:
see attached study protocol

ELIGIBILITY:
Inclusion criteria for people with head and neck cancer:

* minimal age 18
* diagnosis of a primary head and neck squamous cell carcinoma within the last 24 months
* oral, pharyngeal, or laryngeal cancer stage III or IV
* completed surgery and/or radio(chemo)therapy in curative intent

Exclusion criteria for people with head and neck cancer:

* not having the physical, mental, and cognitive ability to understand, follow and hold a conversation in (Swiss-)German
* treatment in palliative intent
* recurrence of the head and neck tumour (local or distant)

Inclusion criteria for significant others of people with head and neck cancer:

* minimal age 18
* being a significant other (partner, spouse, close family member or friend) of an individual with a head and neck cancer with the above-mentioned criteria
* having the permission of the individual affected by head and neck cancer to talk about their experiences

Exclusion criteria for significant others of people with head and neck cancer:

- not having the physical, mental, and cognitive ability to understand, follow and take part in a group discussion in (Swiss-)German

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: individual interview participants: 12 individuals with a diagnosis of a stage III or IV head and neck squamous cell carcinoma, after surgery & (chemo)radiotherapy
  focus group interview participants: 8 significant others (partner, spouse, close familiy member or friend) of individuals with a diagnosis of a stage III or IV head and neck squamous cell carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-03-30 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
interview transcripts | March 2024- May 2025
  individual interviews and focus group interviews will be transcribed verbatim to be analyzed

SECONDARY OUTCOMES:
personal information of participants | March 2024- May 2025
  characteristics of interview and focus group participants will be collected to be able to describe the study participants, including age, education level, cancer stage, treatment received, activity levels

CONTACTS AND LOCATIONS:
Overall Officials: Martina Schmocker, MSc, Principal Investigator — Cantonal Hospital Winterthur, Switzerland
Locations (1):
- Kantonsspital Winterthur, Winterthur, Canton of Zurich, Switzerland

DOCUMENTS (1):
  • Study Protocol (2025-03-28): https://cdn.clinicaltrials.gov/large-docs/13/NCT06272513/Prot_001.pdf